CLINICAL TRIAL: NCT03039348
Title: Keuze Voor Wel of Geen Borstreconstructie na Mastectomie: Onderzoek Naar beïnvloedende Factoren
Brief Title: Opting for Breast Reconstruction After Mastectomy or Not: Search for Influencing Factors
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Principal Investigator, Laura Mettepenningen, student, Universitair Ziekenhuis Brussel
Other Study IDs: v2.0-11/01/2017-LauraM
Record Dates: First submitted 2016-12-11; First posted 2017-02-01 (Estimated); Last update posted 2017-02-01 (Estimated); Status verified 2017-01

CONDITIONS: Breast Cancer Female; Mastectomy; Breast Reconstruction
Keywords: Breast Cancer Female; Mastectomy; Breast Reconstruction; questionnaire

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Breast reconstruction: The patients choosing for breast reconstruction after mastectomy for breast cancer.
  Interventions: Other: semi-structured interview using a questionnaire
- No breast reconstruction: The patients not choosing breast reconstruction after mastectomy for breast cancer.
  Interventions: Other: semi-structured interview using a questionnaire

INTERVENTIONS:
Other: semi-structured interview using a questionnaire — semi-structured interview using a questionnaire

SUMMARY:
The purpose of this study is to investigate the factors influencing the decision about breast reconstruction after breast amputation for breast cancer.

The study will be conducted at the University Hospital in Brussels using only a questionnaire. The results might help us to evaluate and improve the satisfaction among patients about the received information and guidance.

DETAILED DESCRIPTION:
The questionnaire will be completed during one interview. This interview will take place preferably right after the patient visited her doctor at the Breast Clinic at the University Hospital in Brussels.

Before starting the interview all the necessary information to decide whether or not to participate in the study will be given as well as the time to read the informed consent carefully.

ELIGIBILITY:
Inclusion Criteria:

* female
* Dutch speaking
* must have undergone a mastectomy for breast cancer in the following period: 2010 - 2015
* must be a patient of the Breast Clinic at the University Hospital in Brussels

Exclusion Criteria:

* bilateral preventive mastectomy (and therefore no history of breast cancer in any of the breasts)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients of the Breast Clinic at the University Hospital in Brussels.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2016-12; Primary Completion 2017-05 (Estimated); Study Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
factors influencing the choice concerning breast reconstruction after mastectomy, assessed with a questionnaire (with multiple choice and open questions) | december 2016 - may 2017

CONTACTS AND LOCATIONS:
Overall Officials: Laura Mettepenningen, Principal Investigator — Universitair Ziekenhuis Brussel

IPD SHARING:
Plan to Share IPD: Undecided
undecided

REFERENCES:
- [Background] Ananian P, Houvenaeghel G, Protiere C, Rouanet P, Arnaud S, Moatti JP, Tallet A, Braud AC, Julian-Reynier C. Determinants of patients' choice of reconstruction with mastectomy for primary breast cancer. Ann Surg Oncol. 2004 Aug;11(8):762-71. doi: 10.1245/ASO.2004.11.027. Epub 2004 Jul 12. PMID 15249342
- [Background] Fallbjork U, Karlsson S, Salander P, Rasmussen BH. Differences between women who have and have not undergone breast reconstruction after mastectomy due to breast cancer. Acta Oncol. 2010;49(2):174-9. doi: 10.3109/02841860903490069. PMID 20100155
- [Background] Duggal CS, Metcalfe D, Sackeyfio R, Carlson GW, Losken A. Patient motivations for choosing postmastectomy breast reconstruction. Ann Plast Surg. 2013 May;70(5):574-80. doi: 10.1097/SAP.0b013e3182851052. PMID 23542859
- [Background] Gopie JP, Hilhorst MT, Kleijne A, Timman R, Menke-Pluymers MB, Hofer SO, Mureau MA, Tibben A. Women's motives to opt for either implant or DIEP-flap breast reconstruction. J Plast Reconstr Aesthet Surg. 2011 Aug;64(8):1062-7. doi: 10.1016/j.bjps.2011.03.030. Epub 2011 Apr 22. PMID 21514261